CLINICAL TRIAL: NCT01830192
Title: REM (Risk Of Endometrial Malignancy): A Proposal for a New Scoring System to Evaluate Risk of Endometrial Malignancy
Brief Title: REM (Risk Of Endometrial Malignancy)
Acronym: REM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Roberto Angioli, Professor, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 47/09 RA CBM; NCT01830179 (obsolete NCT alias)
Record Dates: First submitted 2013-04-05; First posted 2013-04-12 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Endometrial Disease
Keywords: endometrial cancer; score; nomogram; ultrasound; HE4
MeSH Terms: conditions — Uterine Diseases; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training set (Other): We evaluate the clinical, ultrasound and laboratory features to predict endometrial cancer disease preoperative
  Interventions: Other: Training set
- VERIFICATION SET (Other): We evaluate the clinical, ultrasound and laboratory features to predict endometrial cancer disease preoperative
  Interventions: Other: VERIFICATION SET

INTERVENTIONS:
Other: Training set — We evaluate the clinical, ultrasound and laboratory features to predict endometrial cancer disease preoperative
  Arms: Training set
Other: VERIFICATION SET — We evaluate the clinical, ultrasound and laboratory features to predict endometrial cancer disease preoperative
  Arms: VERIFICATION SET

SUMMARY:
The purpose of this study was to obtain a predictive model to asses the Risk of Endometrial Malignancy (REM) in women with ultrasound endometrial abnormalities.

DETAILED DESCRIPTION:
Objective: It is often difficult to distinguish a benign endometrial disease from a malignancy and tools to help physician are needed, in order to triage patients into high and low risk of endometrial cancer (EC). The purpose of this study was to obtain a predictive model to asses the Risk of Endometrial Malignancy (REM) in women with ultrasound endometrial abnormalities.Women, between 45 and 80 years, diagnosed with ultrasound endometrial abnormalities and scheduled to have surgery were enrolled on a prospective study at Department of Gynaecologic Oncology of Campus Bio-Medico of Rome. Preoperative clinical, ultrasound and laboratory features were taken into account. Logistic regression algorithm was utilized to categorize patients into low and high risk groups for EC.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 45 and 80 years;
2. Eastern Cooperative Oncology Group performance status 0-2 according to World Health Organization (WHO) criteria;
3. informed consent obtained from the patients.

Exclusion Criteria:

1. abnormal cardiac, haematological, renal, respiratory and/or hepatic functions;
2. presence of a previous malignancy;
3. presence of concomitant adnexal masses.

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 741 (Actual)
Dates: Start 2010-01; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
REM (RISK OF ENDOMETRIAL MALIGNANCY): a proposal for a new scoring system to evaluate risk of endometrial malignancy. | 2 year
  We select patients affected by endometrial cancer and benign endometrial disease. Preoperative they underwent to pelvic ultrasound, CA125 and HE4 dosage and anamnesis. They will be considered as training group to obtaine the probability of endometrial malignancy based on HE4, ultrasound features and symptoms.

SECONDARY OUTCOMES:
REM | 2 years
  We select a verification set, composed by endometrial cancer disease and benign endometrial pathologies patients. In this set we apply the risk of endometrial cancer tool, obtained in the training set, in order to verify the sensitivity, specificity and reproducibility.

OTHER OUTCOMES:
REM | 2 years
  We consider training and verification set together to evaluate the overall sensitivity and specificity of predictive tool

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Angioli, MD, Principal Investigator — Campus Biomedico University of Rome
Locations (1):
- campus bio-medico of Rome, Rome, Italy